CLINICAL TRIAL: NCT02109250
Title: CAPRELSA® REGISTRY: a Belgian Registry to Evaluate the Use of Vandetanib (Caprelsa®) in Current Clinical Practice
Acronym: CaprelsaReg
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: D4200R00001
Record Dates: First submitted 2014-03-27; First posted 2014-04-09 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Medullary Thyroid Cancer
Keywords: Medullary Thyroid Cancer (MTC) vandetanib caprelsa
MeSH Terms: conditions — Carcinoma, Medullary | interventions — vandetanib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all Belgian patients treated with Caprelsa® (vandetanib): It is planned to include all Belgian patients diagnosed with aggressive and symptomatic unresectable locally advanced or metastatic Medullary Thyroid Cancer (MTC) who have been prescribed Caprelsa® (vandetanib).
  Interventions: Drug: Caprelsa

INTERVENTIONS:
Drug: Caprelsa — Caprelsa® 100 mg or 300 mg film-coated oral tablets. Each film-coated tablet contains 100 mg or 300 mg of vandetanib.

SUMMARY:
In this registry it is planned to include all Belgian patients diagnosed with aggressive and symptomatic unresectable locally advanced or metastatic Medullary Thyroid Cancer (MTC) who have been prescribed Caprelsa® (vandetanib).

The characteristics of patients receiving Caprelsa® (vandetanib) will be described. Therefore real life data regarding demographic characteristics, evolution of the disease, RET mutation status, the treatment before, during and after vandetanib, dose and duration of treatment with Caprelsa® (vandetanib) and time of progression or death (if applicable) will be included.

ELIGIBILITY:
Inclusion criteria

The subject population that will be observed in this registry, must fulfil all of the following criteria:

1. Provision of subject Informed Consent
2. Patients diagnosed with aggressive and symptomatic unresectable locally advanced or metastatic MTC
3. Patients who already received a prescription for vandetanib in accordance with the scientific leaflet and fulfilling the reimbursement criteria of vandetanib and who are currently treated or have been treated with vandetanib 100 mg or 300 mg tablets.

The prescription of the medicinal product is clearly separated from the decision to include the subject in the registry.

Exclusion criteria Not applicable since patients participating in another study can take part in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include all Belgian sites which have patients diagnosed with aggressive and symptomatic unresectable locally advanced or metastatic MTC who have been prescribed vandetanib and fulfilling the criteria for reimbursement.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this registry is to describe the characteristics of patients who receive Caprelsa® and who are fulfilling the reimbursement criteria. | Up to 16 months
  In this registry the following real life data will be collected: demographic characteristics, evolution of the disease, RET mutation status, the treatment before, during and after vandetanib, dose and duration of treatment with vandetanib and time of progression or death (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Belgium (8):
  - Clinique du Sud Luxembourg, Arlon
  - AZ Klina, Brasschaat
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - UCL St-Luc, Brussels
  - UZ Gent, Ghent
  - AZ Delta, Roeselare
  - CH de Wallonie, Tournai

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2940&filename=8-P102-cv-CT12_NIS_PrimaryReport_CaprelsaRegistry_final_29.09.2015SYNOPSIS_TCC.pdf